CLINICAL TRIAL: NCT06868875
Title: Data Sharing With Collaborative Partners to Develop Computer Aided Detection for the Assessment of the Small Bowel Using MRI
Brief Title: Anonymous Data Sharing for Small Bowel
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 66975
Record Dates: First submitted 2025-02-20; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Small Bowel Disease; Gastrointestinal Diseases
Keywords: Observational
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anonymised datasets acquired as part of an ethically approved research project 'RESEARCH DATASETS':: We have two ongoing ethically approved UCLH studies investigating the use of MRI in small bowel Crohn's disease and comparison with clinical standards of reference, notably endoscopic biopsy, blood test data and clinical symptom diaries. As part of these projects, patients agree to their anonymised data to be used for future work.
  Only staff on the delegation log for the original research project will have access to any psudeo-anonymised datasets acquired as part of that research. This is consistent with ICH Good Clinical Practice and local Research Governance procedures.
- Anonymised datasets acquired as part of clinical practice 'CLINICAL DATASETS': Many patients undergoing small bowel MRI or USS at UCH and other collaborating hospitals often also undergo additional tests as part of their usual clinical care which are recognised as good standards of reference against which we can validate our imaging findings. Notable examples are blood tests (eg. CRP), endoscopy and biopsy, and symptom questionnaires. Furthermore, many patients have normal examinations and these datasets are also very useful in software development to define a standard of normality.
  Only staff with full or honorary contracts and part of the clinical team at collaborating hospitals will have access to the clinical data and un-anonymised datasets. This is consistent with the situation presently as such staff already can access both the PACS and hospital CDR as part of their usual clinical practice

SUMMARY:
Crohn's disease is characterised by an abnormal immunological response within the bowel wall leading to abnormal wall thickening, stricturing (narrowing), fistulation (abnormal connections) to adjacent organs and strictures (narrowing), abnormal motility, and local sepsis (infection). Radiological imaging of the small bowel defines diagnosis, disease extent, biological activity and complications and is vital for timely and efficacious clinical management. Small bowel magnetic resonance imaging (MRI) does not impart ionising radiation and is proving to be a safe, well tolerated and robust method of assessing the small bowel and is widely implemented in the NHS and Europe. MRI evaluates multiple disease related features such as bowel wall thickness and motility which are proving increasing reliable for disease identification, staging, therapeutic guidance and assessment of treatment response.

Currently however radiologists must manually make these measurements which are time consuming and difficult.

There are no computer tools that can quickly and accurate make relevant measurements on MRI to guide patient management. Radiologists at University College Hospital have formed collaborations with groups within University College London (UCL) and around Europe. The investigators have received grant funding to develop computer software to accurately assess the small bowel using MRI over 3 years. To develop this software, it is necessary to use anonymised datasets from patients with and without Crohn's disease undergoing small bowel MRI. Part of this project will require prospective collection of MRI data which has been granted ethical approval as a major amendment to a currently running project (09/H0714/62). The department of Radiology at UCLH has been running a clinical small bowel MRI service since 2005 and have several hundred datasets on its PACS. This current ethics application seeks permission to datashare with the collaborative partners fully anonymised MRI datasets and relevant clinical data from patients previously undergoing small bowel MRI for clinical indications at UCLH.

DETAILED DESCRIPTION:
The investigators wish to share with collaborative partners selected fully anonymized MRI datasets and associated relevant clinical data (such as blood tests results, endoscopic findings, histology) acquired as part of routine clinical practice at UCH since 2005.

The collaborative partners are:

1. The Centre for Medical Image Computing (CMIC) at UCL
2. A European consortium (including UCL as partner and UCLH as subcontractor) which has been awarded an FP7 European grant: University of Delph, Amsterdam medical centre, Eldgenössische Technische Hochschule Zürich, Switzerland, Zuse Institut Berlin, Germany, Biotronics3D Limited UK and Vodera Limited UK.

The investigators wish to share a total of 75 datasets with the FP7 consortium and 300 with CMIC.

Process for the sharing of anonymized datasets acquired as part of clinical practice.

Many patients undergoing small bowel MRI at UCH often also undergo additional tests as part of their usual clinical care which are recognized as good standards of reference against which the investigators can validate our MRI findings. Notable examples are blood tests (eg CRP), and endoscopy and biopsy. Furthermore, many patients have normal examinations and these datasets are also very useful in software development to define a standard of normality.

Suitable datasets will be found as follows:

1. Search of the PACS database to identify all small bowel examinations performed at UCH
2. Use clinical sources freely available to hospital clinical staff via the CDR web system at UCH to triage these patients into relevant clinical groups notably those who have normal small bowel examinations, and those with abnormal studies who have a relevant clinical standard of reference performed within 6 weeks (CRP level, endoscopy, biopsy)
3. Select a sample of relevant datasets for use in software development. The total number to be data shared with the FP7 consortium listed above will not exceed 75. The total number of datasets to be data shared with UCL (CMIC) will not exceed 300. The larger number shared with CMIC reflects their need for a large database of normal examinations to develop motility software.

ELIGIBILITY:
Inclusion Criteria:

* Had a small bowel MRI at UCLH between 2005 and Sept 2010 as part of routine clinical practice who:
* Have a clinical standard of reference within 6 weeks of the MRI scan
* Patients with normal small bowel MRI studies and no clinical evidence of bowel pathology on any additional diagnostic investigations

Exclusion Criteria:

* Patients <16 or not fulfilling either inclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anonymised datasets acquired as part of an ethically approved research project 'RESEARCH DATASETS':
  The investigators have two ongoing ethically approved UCLH studies investigating the use of MRI in small bowel Crohn's disease and comparison with clinical standards of reference, notably endoscopic biopsy, blood test data and clinical symptom diaries. As part of these projects, patients agree to their anonymised data to be used for future work.
  Anonymised datasets acquired as part of clinical practice 'CLINICAL DATASETS':
  Many patients undergoing small bowel MRI or USS at UCH and other collaborating hospitals often also undergo additional tests as part of the usual clinical care which are recognised as good standards of reference against which the investigators can validate their imaging findings.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-04-24 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Develop computer software to extract the bowel from the MRI dataset | Through study completion, an average of 10 years
  measure parameters which reflect Crohn's disease activity which will be used to create and validate models of those parameters which best reflect disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Taylor, Principal Investigator — University College, London
Locations (1):
- University College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT06868875/Prot_SAP_000.pdf